CLINICAL TRIAL: NCT06090604
Title: Movement Amplification Training to Enhance Walking Balance Post-Stroke
Brief Title: Walking Balance Training Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD112813-01 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-10-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Balance control; Walking dysfunction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control of lateral COM motion during and after walking practiced in the MAE (Experimental): For Aim 1a, participant's preferred and fast treadmill walking speeds will be determined followed by 2-min of baseline walking. Each participant will perform eight 2-min trials of treadmill walking 1) Null Environment: no forces, 2) MAE Low Gain: 25 Nsm-1, 3) MAE Medium Gain: 35 Nsm-1, 4) MAE High Gain: 45 Nsm-1, that will be repeated at both treadmill walking speeds. The trial order will be randomized.
  For Aim 1b, we will assess participant's maximum ability to control their lateral COM motion with no forces applied, using three 21-meter walking trials with visual projections on the treadmill to provide feedback used to challenge their lateral COM motion control. Five 2-min trials in a Null environment will be followed by COM control assessment. Participants will rest and repeat the above sequence in a MAE. The order of the external environments will be randomized across participants.
  Participants may participate in more than one aim (1a, 1b and 2).
  Interventions: Other: High intensity gait training in a balance challenging Movement amplification environment

INTERVENTIONS:
Other: High intensity gait training in a balance challenging Movement amplification environment — For Aim 2, each participant will engage in ten 45-min high-intensity gait training sessions performed in a Movement Amplification Environment (MAE). Training sessions will occur 2x/week and led by a licensed Physical Therapist. The goal of each training session is to achieve 40-min of stepping practice within a targeted range of heart rate (HR) of 70 to 80% of estimated age-predicted HR max and perceived excursion (RPE) in a MAE. Each session will begin and end with a 2.5-min warm-up and cool down, with 40-min of training using two 10-min Speed-training blocks and two 10-min Balance-training blocks. Balance training activities will include lateral maneuvers, head turns, obstacle negotiation, and backward walking. The MAE gain, training speeds and balance activities will be progressively increased within and across sessions to challenge the participant.

SUMMARY:
Stroke is one of the leading causes of disability in the United States, affecting ~795,000 people annually. Among ambulatory people with chronic stroke, impaired balance is common and substantially limits mobility (those with the poorest balance walk the least). This project will explore if a novel gait training intervention using a robotic device to amplify a person's self-generated movements can improve walking balance in people with chronic stroke. The development of effective interventions to increase walking balance among people with chronic stroke will positively impact quality of life and ability to participate in walking activities.

DETAILED DESCRIPTION:
Background: People with chronic stroke (PwCS) have substantial walking balance dysfunctions that limit independence and participation in walking activities. There is a pressing need to develop effective methods to enhance walking balance in PwCS. Interventions that amplify self-generated movements may accelerate motor learning by enhance a person's perception of movement errors. This method could potentially be applied to help PwCS improve walking balance. To this end, we have developed a cable-driven robot to create a Movement Amplification Environment (MAE) during treadmill walking. The MAE challenges walking balance by applying lateral forces to the pelvis that are proportional in magnitude to real-time lateral center of mass (COM) velocity. Our purpose is to evaluate effects of MAE training on walking balance in PwCS.

Specific Aims: Aim 1a: To quantify locomotor adaptations PwCS make to maintain walking balance in a MAE. We will evaluate the impact of the two foremost gait training variables: Gait Speed and MAE Strength. Aim 1b: To evaluate short-term changes in the ability of PwCS to control their lateral COM excursion during walking (a quantifiable walking balance measure) immediately after MAE training. Aim 2: To evaluate long-term changes in walking balance and daily walking following a 5-week high-intensity gait training intervention performed in a MAE.

Approach: Aims 1a & b: Twenty PwCS will each participate in two experiments evaluating gait biomechanics (COM dynamics and stepping patterns) during and immediately following MAE training. Aim 1a will evaluate locomotor adaptations when walking in a MAE and the effect of gait speed (slow, preferred, and fast) and MAE strength (low, medium, and high). Aim 1b will use visual feedback to challenge PwCS to control their lateral COM excursion during walking immediately before and after walking in different external conditions (No applied forces, or MAE). Outcomes will assess if short-term walking balance is enhanced immediately following MAE exposure. Aim 2: Ten PwCS will participate in 10-sessions of high intensity gait training performed in a MAE. We will assess pre- to post- changes in walking balance using clinical gait and balance measures, biomechanical assessments, and participation in daily walking (steps/day). Outcomes will assess if long-term walking balance is enhanced following MAE gait training.

Impact: Training walking balance of PwCS by amplifying their own self-generated movements is a radical departure from current practice and could substantially enhance walking balance. This study will provide a foundational understanding of how PwCS maintain walking balance in a MAE and if beneficial behaviors persist following MAE training. Successful outcomes will motivate a randomized controlled trial assessing efficacy of MAE training on walking balance in PwCS.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. diagnosis of hemiparetic stroke;
3. more than 6 months post-stroke;
4. ability to ambulate over ground for 10 meters with or without a single cane, and/or ankle-foot orthosis.

Exclusion Criteria:

1. cognitive impairment (score of ≤22/30 on the Montreal Cognitive Assessment scale);
2. aphasia (score of ≥71/100 on the Mississippi Aphasia Screening Test);
3. excessive spasticity in lower limbs (score of > 3 on the Modified Ashworth Scale);
4. unable to tolerate 10-min. of standing;
5. enrollment in concurrent physical therapy;
6. use of braces/orthotics crossing the knee joint;
7. known pregnancy;
8. severe cardiovascular, musculoskeletal, or other neurological conditions affecting gait and balance.
9. brainstem and/or cerebellar lesion
10. perinatal stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Minimum average lateral center of mass (COM) excursion | For Aim 1, COM excursion will be calculated at session 1 and after a week on session 2. For Aim 2, COM excursion will be calculated at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  Minimum average lateral COM excursion occurring during 5 consecutive gait cycles will be calculated as our metric of ability to control lateral COM motion during walking
Minimum lateral margin of stability | For Aim 1, margin of stability will be calculated at session 1 and after a week on session 2. For Aim 2, margin of stability will be calculated at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  Minimum lateral margin of stability is the distance between the lateral extrapolated center of mass (XCOM) and the base of support (BOS), approximated as the lateral position of the 5th metatarsal marker on the side of the last initial contact. Minimum MOS is identified during stance phase of each step. Extrapolated center of mass (XCOM) position is calculated using:
  XCOM= COM + COM* √ l/g
10 Meter Walk Test (10MWT) | For Aim 1, 10MWT will be performed at session 1 to determine baseline functional status. For Aim 2, 10MWT will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  10MWT is a simple measurement of an individual's average walking speed measured at self-selected speed (instruction: "walk at your normal comfortable pace") and fastest-possible speed (instruction: "as fast as you safely can").
Timed Up and Go (TUG) | For Aim 1, TUG will be performed at session 1 to determine baseline functional status. For Aim 2, TUG will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  TUG is used to assess functional mobility, walking balance, and fall risk. It is a quick, valid, reliable and widely used clinical performance based measure in individuals post-stroke. While there is no time limit to the TUG test, more time taken to finish the task indicates poor balance and greater fall-risk.
Berg Balance Scale (BBS) | For Aim 1, BBS will be performed at session 1 to determine baseline functional status. For Aim 2, BBS will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  BBS is a 14-item measure that assesses static balance with excellent validity and reliability in individuals post-stroke. The total score for this test is 56. Minimum score is 0 and maximum score is 56. Higher scores indicate better balance and lower fall-risk, while lower scores indicate poor balance and increased fall-risk.
Activities-specific Balance Confidence (ABC) Scale | For Aim 1, ABC will be performed at session 1 to determine baseline functional status. For Aim 2, ABC will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  ABC scale is a self-reported measure of an individual's confidence while performing specific postural and ambulatory activities. The ABC is a reliable and valid measure of balance confidence in individuals post-stroke. The total score for ABC scale is 1600. Minimum score is 0 and maximum score is 1600. Higher scores indicate better balance confidence, while lower scores indicate poor balance confidence.
Dynamic Gait Index (DGI) | For Aim 1, DGI will be performed at session 1 to determine baseline functional status. For Aim 2, DGI will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  DGI is an eight item test that assesses gait, balance and fall risk during usual steady-state walking and walking during more challenging tasks. The total score for this test is 24. Minimum score is 0 and maximum score is 24. Higher scores indicate better walking balance, while lower scores indicate poor walking balance.
6 minute walk test (6WMT) | For Aim 2, 6WMT will be performed at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered during 6 minutes of walking indicate participants exercise tolerance. The vitals measures before and after the 6MWT indicate the cardiovascular and respiratory response to exercise.
Stepping Activity in the Home and Community | For Aim 2, the stepping activity will be assessed for a period of one week after session 1 and session 12 (post 5 weeks of training). Participants will be asked to wear the monitor during all waking hours.
  The amount of daily stepping in the home and community taken per day averaged across the 7-day collection periods before and after training will be assessed for Aim 2. Daily stepping will be measured and recorded using a StepWatch4 (Modus, Edmonds, WA) activity monitor. The microprocessor-based accelerometer will be worn around the ankle during all waking hours (except bathing) for the duration of the stepping assessment period.

SECONDARY OUTCOMES:
Step length | For Aim 1, step length will be performed at session 1 and after a week on session 2. For Aim 2, step length will be calculated at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  Step length is calculated as the fore-aft distance between the calcanei markers at initial foot contact.
Step width | For Aim 1, step width will be performed at session 1 and after a week on session 2. For Aim 2, step width will be calculated at session 1 and after 5 weeks of training at session 12. Each of these sessions will be two hours long.
  Step width is calculated as the medio-lateral distance between the left and right 5th Metatarsal markers at initial foot contact
Heart rate | For Aim 2, heart rate will be collected before and after each of the 10 one hour long training sessions over 5 weeks. Vitals will be collected at session 1 and after 5 weeks of training at session 12. Both these sessions will be two hours long.
  Participants heart rate in beats per minute (bpm) will be collected to determine cardiovascular response to exercise.
Blood pressure | For Aim 2, blood pressure will be collected before and after each of the 10 one hour long training sessions over 5 weeks. Vitals will be collected at session 1 and after 5 weeks of training at session 12. Both these sessions will be two hours long.
  Participants blood pressure in millimeters of mercury (mm Hg) will be collected to determine cardiovascular response to exercise.
Exertion | For Aim 2, participants level of exertion will be collected throughout the 10 training sessions over 5 weeks. Each training session will be one hour long.
  Participants exertion monitored via 6-20 point rate of perceived exertion scale and heart rate will be collected to determine participants performance during each training session and track their progress. Minimum score for perceived exertion is 6 and maximum score is 20. Higher score indicates greater exertion and lower score indicates less exertion.
Number of steps taken during training session | For Aim 2, the total number of steps during training will be collected after each of the 10 training session over 5 weeks. Each training session will be one hour long.
  Participants number of steps taken during the training session will be collected to determine participants performance during each training session and track their progress.
Chedoke-McMaster Stroke Assessment (CMSA) scale | For both Aims 1 and 2, CMSA scale will be collected at session 1 to determine participants stroke recovery. This session will be two hours long.
  CMSA will be collected to determine the level of stroke impairment in participants leg and foot. Each domain (leg and foot) are scored on a 7-point scale (stage 1 through 7, most impairment through to no impairment, respectively). Minimum score is 0 and maximum score is 7.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Gordon, PhD, Principal Investigator — Assistant Professor, Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study will be uploaded on the Northwestern University Research and Data repository (Arch) so that it is fully available to other parties interested in probing the data further and performing secondary analyses.
Supporting Information: Study Protocol
Time Frame: After completion of the study
Access Criteria: Data will be publicly available.